CLINICAL TRIAL: NCT02653495
Title: Impact of Metabolic Syndrome on Flu Vaccine Efficacy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Target accrual not met
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UAN-0891
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Results first posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Immune Deficiency; Metabolic Syndrome
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Metabolic Syndrome | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Influenza vaccine in metabolic syndrome (Experimental): Influenza vaccine
  Interventions: Biological: Influenza vaccine
- Influenza vaccine in healthy controls (Experimental): Influenza vaccine
  Interventions: Biological: Influenza vaccine

INTERVENTIONS:
Biological: Influenza vaccine — Influenza vaccine administered intramuscularly (IM), 1 time only, on visit 3

SUMMARY:
Metabolic syndrome (MetS) is a cluster of metabolic conditions associated with obesity that predispose individuals to coronary heart diseases and diabetes but obesity has been shown to increase the risks of other diseases like cancer and asthma. Studies have also shown that obesity increases the risk of severe influenza infection and associated death and reduces the efficacy of influenza vaccine in the obese population but yet, the molecular mechanisms have not been described. The investigators are thus hypothesizing that differences in the innate immune responses between individual with or without metabolic syndrome impact viral infection and vaccine outcome. The investigators will perform seasonal influenza vaccination in people with or without metabolic syndrome to determine if the late adaptive response assessed by antibodies titers is different between the two groups and correlates with the early immune response assessed by gene expression profile in whole blood cells. The project proposed by the investigators will contribute to a better understanding of the inflammatory phenotype associated with metabolic syndrome and establish for the first time if it affects the immune protection against infectious diseases and particularly against influenza virus infection. The results will be important to determine if the population affected by metabolic syndrome should receive anti-influenza treatment in priority in the context of a severe influenza epidemic.

DETAILED DESCRIPTION:
The development of industrialization with increased food consumption and sedentarity has given rise to an obesity pandemic, which affects up to 30% of the population in countries like US, these populations being at greater risk for cardiovascular diseases, and diabetes. More than obesity per se, visceral obesity is associated with metabolic diseases that cluster together and clinically defined metabolic syndrome. MetS comprises individuals with at least three of the 5 of the following factors: abdominal obesity, high blood triglycerides, low HDL ("good cholesterol"), high blood pressure and elevated fasting glucose. Metabolic syndrome is associated with a low-grade inflammation characterized by an infiltration of immune cells particularly in the adipose tissue, the liver and the pancreas that is thought to be responsible for the induction of insulin resistance. It is thought that obesity predisposes to other diseases such as cancer, asthma but only little attention has been given to infectious diseases. Studies have shown that obesity increases the risk of severe influenza infection and associated death and reduces the efficacy of influenza vaccine in the obese population but yet, the molecular mechanisms have not been described. Immune dysfunctions associated with obesity are suspected to play a major role but obesity is often associated with respiratory disorders that could directly explain the increased susceptibility to influenza infection. Also, metabolically healthy obesity is less associated with inflammation. Therefore, the investigators would like to focus particularly on metabolic syndrome, and determine how it influences immune response to viruses.

The investigators are thus hypothesizing that differences in the innate immune responses between individual with or without metabolic syndrome impact viral infection and vaccine outcome. Recent studies involving complex biological analysis and computational modeling have shown that the ability of an individual to positively respond to influenza vaccine can be molecularly predicted by looking at markers in the blood cells. The investigators will perform seasonal influenza vaccination in people with or without metabolic syndrome to determine if the late adaptive response assessed by antibodies titers is different between the two groups and correlates with the early immune response assessed by gene expression profile in whole blood cells.

Healthy nutritional habits along with increased physical activities should be best at preventing the development of metabolic syndrome but socio-economical issues are slowing the implementation of these changes. Therefore, as metabolic syndrome is raising public health concerns, it is important to understand why the metabolic syndrome affects susceptibility to diseases.

ELIGIBILITY:
Inclusion criteria for the METABOLIC SYNDROME COHORT( Participants must have 3 or more of the following 5 risk factors):

* Abdominal Obesity, given as a waist circumference: Men >102 cm (>40 in) Women > 88 cm (>35 in)
* Triglycerides >150 mg/dl
* HDL Cholesterol: Men < 40 mg/dl Women < 50 mg/dl
* Blood Pressure >130/ >85 mm Hg - or controlled on antihypertensive medication
* Fasting Glucose > 100 mg/dl

Inclusion criteria for the HEALTHY CONTROLS (Participants must have all of the requirements below) :

* body mass index 18.5 - 25 kg/m2
* HDL female > 50 mg/dL, male > 40 mg/dL
* fasting glucose < 100 mg/dL
* triglycerides <150 mg/dL,
* waist circumference of a female < 88 cm, male < 102 cm)
* - Blood pressure < or = to 120/80 (based on an average of 3 readings taken 5 minutes apart after the consent form has been signed)

Exclusion criteria :

* Currently undergoing treatment for the metabolic syndrome
* The average of 2 BP readings > 150/90 (based on 2 B/Ps taken at screening visit 1).
* Hepatitis A, B and C
* NSAIDs and/or Aspirin ingestion within the last 14 days
* Self-reported history of any active autoimmune diseases
* Self-reported ingestion of statins within the last 3 months
* Self-reported antibiotic use within the last 3 months
* Anti-inflammatory drugs including biologics and corticosteroids within last 3 months( nasal spray and topical applications are OK)or Omega 3 Fatty Acids.
* Self-reported hx of cancer treatment within the last year
* Allergy to eggs
* History of Guillain-Barre syndrome
* Pregnant ( determined by point of care testing at screening visit 1).
* HIV positive
* Self-reported history of flu vaccination within the past 3 months.
* Any self-reported infection in the week of the visit except the first two visits (Screening visit 1 and Screening visit 2) and the last visit (Study visit #5) that could be rescheduled.
* Any medical, psychological or social condition that, in the opinion of the Investigator, would jeopardize the health or well-being of the participant during any study procedures or the integrity of the data.

Study Population Description The population from which the groups will be selected are resident of New York City.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Andreo, PhD, Principal Investigator — The Rockefeller University Center for Clinical and Translational
Locations (1):
- Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Advertising and Research Volunteer Repository Database
Pre-assignment Details: Pre-screening took place along with a two-step screening visit for eligibility criteria. Those not meeting eligibility would screen out: 86 prescreened, 28 initial contact for screening.
Period: Overall Study
Arm/Group | Influenza Vaccine in Metabolic Syndrome | Influenza Vaccine in Healthy Controls
Started | 15 | 2
Completed | 3 | 2
Not Completed | 12 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Screening Failure | 10 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza Vaccine in Metabolic Syndrome | Influenza Vaccine in Healthy Controls | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Antibody Response D28
Description: Measured by hemagglutination inhibition assay
Time Frame: 28 days after vaccination compare to baseline (screening visit 1) pre-vaccination
Population: Data were not collected
Arm/Group | Influenza Vaccine in Metabolic Syndrome | Influenza Vaccine in Healthy Controls
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Gene Expression Profiling D1
Description: Analyze by RNA-seq
Time Frame: 1 day post-vaccination compare to baseline (gene expression screening visit #1 and study visit #1 D0 of vaccination)
Population: Data were not collected.
Arm/Group | Influenza Vaccine in Metabolic Syndrome | Influenza Vaccine in Healthy Controls
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Gene Expression Profiling D28
Description: Analyze by RNA-seq
Time Frame: 28 days post-vaccination compare to baseline (gene expression screening visit #1 and study visit #1 D0 of vaccination)
Population: Data were not collected.
Arm/Group | Influenza Vaccine in Metabolic Syndrome | Influenza Vaccine in Healthy Controls
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Gene Expression Profiling D90
Description: Analyze by RNA-seq
Time Frame: 90 days post-vaccination compare to baseline (gene expression screening visit #1 and study visit #1 D0 of vaccination)
Population: Data were not collected.
Arm/Group | Influenza Vaccine in Metabolic Syndrome | Influenza Vaccine in Healthy Controls
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Antibody Response D90
Description: Measured by hemagglutination inhibition assay
Time Frame: 90 days after vaccination compare to day 28
Population: Data were not collected.
Arm/Group | Influenza Vaccine in Metabolic Syndrome | Influenza Vaccine in Healthy Controls
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event information collected from time of enrollment through completion of study visits, 3 months.
Arm/Group | Influenza Vaccine in Metabolic Syndrome | Influenza Vaccine in Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/3 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influenza Vaccine in Metabolic Syndrome (N=3) | Influenza Vaccine in Healthy Controls (N=2)
infections and infestations: upper respiratory infection: skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Dog bite on left great toe. Family pet with "all immunizations". Neosporin oint daily and band aid. Ambulatory and comfortable. No redness, swelling, drainage or tenderness. It is healing well.
gastrointestinal disorders: dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) — moderate to severe indigestion after eating brunch. Denies vomiting, diarrhea, sweats or fever. Self treated with pepto bismol with relief. Has history of self-diagnosed gastroesophageal reflux disease (GERD).
gastrointestinal disorders: diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject experienced abdominal cramping and diarrhea after eating food from a street vendor. No fever, no vomiting, was able to eat and drink. Onset 3 days after receiving flu vaccine. Symptoms resolved after 48 hours.
Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Subject called complaining of congestion and cough.

LIMITATIONS AND CAVEATS:
Inclusion Criteria hard to meet among population: many individuals do not self-identify as having metabolic syndrome, participants must have untreated metabolic syndrome. Challenges led to early termination with sample size not being attainable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT02653495/Prot_SAP_000.pdf